CLINICAL TRIAL: NCT03968068
Title: The Effects of Acute Exercise and Remote Ischaemic Conditioning (RIC) on Cerebral Blood Flow Velocity in Patients With Ischaemic Stroke and Healthy Controls
Brief Title: Exercise and RIC and TCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH20750
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Procedure: Exercise Procedure
- Remote Ischaemic Conditioning (Experimental)
  Interventions: Procedure: Remote Ischaemic Conditioning

INTERVENTIONS:
Procedure: Exercise Procedure — Patients will undergo 30 minutes of light-moderate intensity leg cycling, using the Letto-2 (Motomed, UK) in the semi-supine position.
  Arms: Exercise
Procedure: Remote Ischaemic Conditioning — Patients will undergo 4 cycles of upper limb RIC using a blood pressure cuff. Each cycle will involve inflating the blood pressure cuff to 200 mmHg for five minutes around the upper arm, followed by a period of relaxation of the cuff for a further 5 minutes. The total RIC treatment time will take 40 minutes.
  Arms: Remote Ischaemic Conditioning

SUMMARY:
The first week after a stroke is a particularly important time, as improving blood flow may limit secondary ischaemic damage to the brain and help reduce the overall burden neurological injury and future disability.

Small studies in patients with stroke have shown that moderate aerobic exercise increases blood flow to the brain, however, no studies have evaluated the safety of aerobic exercise within the first week after stroke, nor whether it results in changes to cerebral blood flow.

Remote ischaemic conditioning (RIC) is when ischaemia is induced to a limb for short periods of time by inflating pressure cuffs around arms or legs to above systolic pressures (mmHg). This procedure is performed for periods that avoid physical injury to the limbs, but induce neurohormonal, systemic or vascular changes in the body. These changes often result in improved blood supply to various areas of the body. The use of RIC in the acute period after stroke is currently being investigated in a number of large randomised controlled trials e.g. RECAST, RESIST, however, our understanding of how RIC actually works is incomplete. Importantly, there is scarce data on the acute effects of RIC on cerebral blood flow (CBF), a potentially pivotal mechanism behind its effects.

We propose an exploratory study to evaluate whether it is feasible, acceptable and safe to undertake low and moderate intensity aerobic exercise or remote ischaemic conditioning (RIC) in patients during the acute period after stroke, and whether either of these interventions result in changes to cerebral blood flow velocity (CBFv) in the major cerebral arteries. We will compare any changes to those in a cohort of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18) patients who have suffered acute ischaemic stroke between 2-7 days previously, or healthy adult (>18 years).
* Ability to provide written informed consent
* Ability to mobilise lower body limbs (at least one leg)
* Ability to comply with study procedures in the opinion of the treating physician.

Exclusion Criteria:

* Haemorrhagic Stroke
* Ischaemic stroke < 2 days or >10 days
* Disability preventing lower extremity cycling
* New York Heart Failure Classification stage III/IV
* History of ischaemic stroke
* Current diagnosis of cancer
* Resting Blood pressure > 180 / 100 mmHg
* Clinically unstable
* History or presence of significant peripheral vascular disease in the upper limbs.
* History or presence of complex neuropathic pains or peripheral neuropathy in the arms.
* Presence of lymphoedema in the arms.
* Presence of skin ulceration to the arms.
* Uncontrolled arrhythmia, hypertension, diabetes or angina.
* Acute deep vein thrombosis, pulmonary embolism or pulmonary infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Incidences of RICTreatment-Emergent Adverse Events. | 48 hours
  Safety of the RIC intervention will be assessed by measuring the Number of Adverse Events experienced by participants that are related to the RIC intervention.
Number of Incidences of Exercise Treatment-Emergent Adverse Events. | 48 hours
  Safety of the exercise intervention will be assessed by measuring the Number of Adverse Events experienced by participants that are related to the exercise intervention.
Number of participants reporting RIC associated discomfort on a likert scale | 48 hours
  Reported grade of discomfort associated with RIC will be measured on a likert scale of 0-5, 1 being very uncomfortable to 5 being very comfortable. Acceptance of RIC will be defined as an average score of >3/5 on the likert scale.
Number of participants reporting exercise associated discomfort on a likert scale | 48 hours
  Reported grade of discomfort associated with exercise will be measured on a likert scale of 0-5, 1 being very uncomfortable to 5 being very comfortable. Acceptance of exercise will be defined as an average score of >3/5 on the likert scale.
% of RIC intervention completed and recorded | 48 hours
  Feasibility of RIC will be defined as >80% of the intervention being completed and recorded.
% of exercise intervention completed and recorded | 48 hours
  Feasibility of exercise will be defined as >80% of the intervention being completed and recorded.

SECONDARY OUTCOMES:
Change from baseline in cerebral blood flow velocity. | 48 hours
  Cerebral blood flow velocity will be measured using Transcranial Doppler (TCD).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ali, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided